CLINICAL TRIAL: NCT05616585
Title: Dietary Biomarkers Development Center at Harvard University: Intervention Core
Brief Title: Dietary Biomarkers Intervention Core
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Frank Sacks, Principal Investigator, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB21-1067; 1U2CDK129670-01 (NIH)
Record Dates: First submitted 2022-10-28; First posted 2022-11-15 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Biological Markers; Diet, Healthy; Metabolomics; Nutrition, Healthy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharmacokinetic (Experimental): Single Day Intervention of 10 test foods
  Interventions: Other: Pharmacokinetic (PK)- Controlled Feeding Diet
- Dose Response (Experimental): Six day, 3 level (zero, medium, high dose) controlled feeding study
  Interventions: Other: Dose Response (DR)- Controlled Feeding Diet

INTERVENTIONS:
Other: Pharmacokinetic (PK)- Controlled Feeding Diet — Pharmacokinetic- single-day isocaloric meals of beef, potatoes, chicken, whole wheat bread, corn, cheese, yogurt, and oats with blood and urine samples taken at Time Zero and every hour (blood) or two hours (urine) after eating, over 10 hours; and at 24 hr.
  Arms: Pharmacokinetic
Other: Dose Response (DR)- Controlled Feeding Diet — Dose Response-3 level, six days controlled feeding study with assignment to either beef/whole wheat bread, chicken/potato, salmon/corn, cheese/soybeans, or yogurt/oats within a standard diet at zero, medium, and high doses for 6 days.
  Arms: Dose Response

SUMMARY:
The purpose of this controlled feeding trial is to establish an Intervention Core, equipped to perform tightly controlled pharmacokinetic (PK) and dose-response (DR) feeding studies.

This research is a two-component pharmacokinetic and pharmacodynamic cross-over dietary feeding trial.

* In the PK study, eight foods will be tested, each on a single day, and the design is crossover.
* In the DR, the effects of 10 foods will be compared to each other in a randomized, parallel-group design, and the dose-effect of each of the 10 foods will be determined in a randomized, crossover design.

DETAILED DESCRIPTION:
Diet is one of the most important determinants of human health and an essential component of population-wide primary prevention strategies. However, there is controversy about the quality and reliability of population- based nutrition research. The vast majority of evidence for healthy eating is informed by large studies with dietary patterns assessed via self-report. Self-reported tools have well-recognized limitations. Plasma biomarkers have been a mainstay of epidemiologic studies. Recent advances in metabolomics technology have similarly fostered discovery of metabolites that are highly specific to intakes of foods or food groups. Metabolomics offers a tangible opportunity to identify novel metabolomic signatures for a range of foods and nutrients. However, this progress relies on the tremendous need for controlled feeding studies to identify and validate metabolites specific to each food item and group.

This research will identify objective biomarkers of dietary intake that can serve as independent markers of dietary intake and complement current dietary intake assessment methods. The knowledge gained in this approach will thus address a critical gap with immediate benefits to the larger nutrition research community, both in observational and clinical trial settings, to improve the validity of major public health research initiatives. The Intervention Core, will perform tightly controlled pharmacokinetic (PK) and dose-response (DR) feeding studies across a range of food items and food groups in diverse populations. The investigators will focus on common foods from the protein, carbohydrates, and dairy food groups: (1) chicken, beef, salmon, and soybeans;(2) yogurt, cheese; and (3) whole wheat bread, potatoes, corn, and oats.

Pharmacokinetic (PK): Each participant will complete a sequence of dietary intakes of up to 8 test foods in a randomized, crossover study, blinded according to the order of randomization. In each of the eight feeding cycles a control diet is provided for a 2 day run-in, after which each participant will be given a pre-specified amount of the test foods, i.e., beef, potatoes, chicken, whole wheat bread, corn, cheese, yogurt, or oats. Blood and urine samples will be taken at time zero, every hour for blood or two hours for urine after eating, over 10 hours, and at 24 hours for untargeted Liquid chromatography-mass spectrometry (LC-MS) metabolomic analysis.

Dose Response (DR):The DR study is an isocaloric, controlled feeding study that will examine three dose levels for 10 foods in five pairings. A total of 100 eligible adults (20 per food group pairing) (will be assigned to beef/potatoes, chicken/whole wheat bread, salmon/corn, cheese/soybeans, or yogurt/oats within a standard diet at zero, medium, and high doses for six days each in a randomized crossover design.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults Men and women, 18+
* Body Mass Index (BMI) 18.5-39.9 kg/m2
* Willingness to participate in all study visits

Exclusion Criteria:

* History of gastrointestinal conditions (e.g., ulcerative colitis, Crohn disease, celiac sprue, Hereditary Non-polyposis Colorectal Cancer, familial adenomatous polyposis, pancreatic disease, liver disease)
* Bleeding disorders that preclude blood draws
* Anemia- as self-reported in the Screening Questionnaire
* Previous gastrointestinal resection or gastric bypass surgery
* Recent hospital admissions (in past 6 months) for heart disease (myocardial infarction, cerebrovascular accident, or congestive heart failure) or other cerebrovascular/ coronary artery disease condition under physician guided therapy that is not medically stable.
* Cancer under radiation or chemotherapy treatment that is active or within 6 months of treatment. Except for non-melanoma skin cancer.
* Women who are pregnant or lactating
* Weight change (±5% in3 months)
* Regular alcohol intake of >2 drinks/day (2 drinks being equivalent to 720 ml beer, 240 ml wine, or 90 ml spirits) and unwilling to abstain during feeding periods
* Use of tobacco, marijuana, hookahs, vape, or e-cigarettes and not willing to abstain during feeding periods.
* Use of illicit drugs and not willing abstain during feeding periods.
* Body mass index >40 kg/m2
* Hypertension- seated blood pressure >140 mmHg or diastolic >90 mmHg
* Food allergies/intolerances or major dislikes to foods used in the study menus; unwilling to consume study foods.
* Regular (daily to weekly) use of over-the-counter weight-loss aids, anti-inflammatories, and unwilling to stop taking these during feeding periods
* Unwilling to stop taking over the counter dietary supplements that interfere with the test foods being studied, including pills, chewable, liquids or powders for the following: protein supplements, soy, fiber, flaxseed, fish oil (incl. cod liver oil), probiotics, carotenoids, selenium, other antioxidants, other phytochemicals, glucosamine, and chondroitin. If vitamin supplement is MD prescribed, the participant may be enrolled subject to the investigator's judgment. Staff will review supplement to determine eligibility.
* Oral or IV antibiotic use in the past 3 months (could defer participation until 3 months post completion of course of antibiotics)
* Inability to freely give informed consent
* Clinical lab tests outside acceptable value as ascertained at a screening blood draw and current use of specific prescription medications per self-report

Description [Acceptable Values]

Glucose-Fasting: Serum Glucose [54-125 mg/dl]

Blood Urea Nitrogen [6-50mg/dl]

Serum Creatinine [0.4-1.3 mg/dl]

Estimated glomerular filtration rate (eGFR) [>60ml/min]

Serum Sodium [133-146 mmol/L]

Alanine Aminotransferase/glutamate-pyruvate transaminase (ALT/GPT) Liver Enzyme [5-60 U/L]

Aspartate aminotransferase (AST/GOT) Liver Enzyme [5-40 U/L]

Alkaline Phosphatase Liver Enzyme [20-135 U/L]

Total Bilirubin Liver Function [0.0-1.9 mg/dl]

Total Serum Protein [5-9.0 g/dl]

Albumin Serum Protein [3.5-5.9 g/dl]

LDL Cholesterol [<160 mg/dl]

Triglycerides [<500 mg/dl]

White Blood Cells (WBC) [3-10.5 K/per microliter (μL)]

Hematocrit (HCT) (women) [35-48 g/dl]

Hematocrit (HCT) (men) [37.5-49 g/dl]

Prescription Medications that would Exclude Participation:

* Diuretics
* Steroids (oral): daily oral any dose within 1 month of study, except as noted below
* Nonsteroidal anti-inflammatory drugs (NSAIDS): when prescribed for treatment or is regularly consumed (i.e.. Daily), or can't be stopped for 2 days without pain, except 81 mg Aspirin
* Opiates: any use within 1 month of study
* Antilipemic Agents that affect GI or renal function (i.e.. Fibrates)
* Antidiabetics and Hypoglycemic medications other than metformin (i.e.. insulin, SGLT2 inhibitor, α-glucosidase inhibitor)
* Psychiatric that affect metabolism/renal function (anti-psychotics, lithium)
* Biologics/immune modulators (i.e.. rheumatoid arthritis (RA), psoriasis, other rheumatologic/hematologic active disease)
* Anti-coagulants (coumadin, heparin, Eliquis, etc.)
* Human immunodeficiency virus (HIV) or highly active antiretroviral therapy (HAART) , etc.

  * Medications that are approved: Steroids (nasal or topical), Aspirin, NSAIDS and Tylenol (avoid day before and day of study visit, Statins, Metformin, Psychiatric drugs other than anti-psychotics (SSRI, tricyclics, benzo), oral contraception pill (OCP)/Hormonal Replacement Therapy (HRT), Tobacco cessation products (patches/lozenge), Oral contraceptives, Gender- affirming HRT, Testosterone for hypogonadal males.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Urinary biomarker changes following consumption of specific foods will be measured using metabolomic approaches in post consumption samples. | Pharmacokinetic Phase1: [Time Frame: 0, 2, 4, 6, 8, 10 and 24 hours post consumption of the test food.] Dose Response Phase 2: [Time Frame: Day 0 and Day 7 post consumption of 6 days controlled feeding of paired test foods.
  Urine samples are taken at baseline and postprandially to determine how the biomarkers behave post consumption, which is standard practice in dietary biomarker identification studies.
  A number of biomarkers will be identified for the test foods. These biomarkers will be measured using liquid chromatography-mass spectrometry (LC/MS) and nuclear magnetic resonance (NMR) spectroscopy and will be reported in relative units. An untargeted approach will be applied to measure the biomarkers, of which hundreds will be measured. These biomarkers will be from different classes of compounds such as amino acids, fatty acids, lipids, and carbohydrates for example. Note: A list of biomarkers has not been added as the investigators are using an untargeted metabolomics approach, which will be used to identify biomarkers from different compound classes.
Serum/plasma biomarker changes following consumption of specific foods will be measured using metabolomic approaches in post consumption samples. | Pharmacokinetic Phase 1 [ Time Frame: 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10 and 24 hours post consumption of the test food.] Dose Response Phase 2: [Time Frame: Day 0 and Day 7 post consumption of 6 days-controlled feeding of paired test foods.
  Blood samples are taken at baseline and postprandially to determine how the biomarkers behave post consumption, which is standard practice in dietary biomarker identification studies.
  A number of biomarkers will be identified for the test foods. These biomarkers will be measured using LC/MS and NMR spectroscopy and will be reported in relative units. An untargeted approach will be applied to measure the biomarkers, of which hundreds will be measured. These biomarkers will be from different classes of compounds such as amino acids, fatty acids, lipids and carbohydrates for example. Note: A list of biomarkers has not been added as the investigators are using an untargeted metabolomics approach, which will be used to identify biomarkers from different compound classes.
Stool biomarker changes following consumption of specific foods will be measured using metabolomic approaches in post consumption samples. | Dose Response Phase 2: [Time Frame: Day 0 and Day 7 post consumption of 6 days-controlled feeding of paired test foods.
  . Stool samples are taken at baseline and postprandially to determine how the biomarkers behave post consumption, which is standard practice in dietary biomarker identification studies.
  A number of biomarkers will be identified for the test foods. These biomarkers will be measured using LC/MS and NMR spectroscopy and will be reported in relative units. An untargeted approach will be applied to measure the biomarkers, of which hundreds will be measured. These biomarkers will be from different classes of compounds such as amino acids, fatty acids, lipids and carbohydrates for example. Note: A list of biomarkers has not been added as the investigators are using an untargeted metabolomics approach, which will be used to identify biomarkers from different compound classes.

CONTACTS AND LOCATIONS:
Overall Officials: Frank M Sacks, MD, Principal Investigator — Harvard School of Public Health (HSPH); Jonathan S Williams, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Mass General Brigham Center for Clinical Investigation, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Chakraborty H, Sun Q, Bhupathiraju SN, Schenk JM, Mishchuk DO, Bain JR, He X, Sun J, Harnly J, Simmons W, Raftery D, Liang L, Newman JW, Fiehn O, Clish CB, Lampe JW, Bennett BJ, Navarro SL, Wang Y, Zheng C, Mossavar-Rahmani Y, McCullough ML, Huang Y, Shojaie A, Zhu W, Djukovic D, Sacks F, Williams J, Steinberg FM, Adams SH, Hu FB, Neuhouser ML, Slupsky CM, Maruvada P. The Dietary Biomarkers Development Consortium: An Initiative for Discovery and Validation of Dietary Biomarkers for Precision Nutrition. Curr Dev Nutr. 2025 Apr 5;9(5):107435. doi: 10.1016/j.cdnut.2025.107435. eCollection 2025 May. PMID 40641655
- See also: Harvard Dietary Biomarkers Website — https://www.hsph.harvard.edu/eat-biomarkers/
- See also: Biomarkers Consortium Website — https://dietarybiomarkerconsortium.org/

DOCUMENTS (2):
  • Informed Consent Form: Dietary Biomarkers Phase 1 Pharmacokinetic (2023-10-06): https://cdn.clinicaltrials.gov/large-docs/85/NCT05616585/ICF_000.pdf
  • Informed Consent Form: Dietary Biomarkers Phase 2 Dose Response (2024-09-11): https://cdn.clinicaltrials.gov/large-docs/85/NCT05616585/ICF_001.pdf